CLINICAL TRIAL: NCT04936893
Title: Effects of Mindfulness Practice on Healthcare Workers During the COVID-19 (Coronavirus Disease) Pandemic
Brief Title: Effects of Mindfulness Practice on Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YaleNUS
Record Dates: First submitted 2021-06-07; First posted 2021-06-23 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Psychological Burnout
MeSH Terms: conditions — Burnout, Psychological | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeadSpace Mobile App (Experimental): Mindfulness practice
  Interventions: Behavioral: Mindfulness Practice
- Lumosity Mobile App (Active Comparator): Cognitive games
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Mindfulness Practice — 10-15 mins of daily mindfulness practice using HeadSpace, for 3 weeks
  Arms: HeadSpace Mobile App
Behavioral: Cognitive training — 10-15 mins of cognitive games using Lumosity, for 3 weeks
  Arms: Lumosity Mobile App

SUMMARY:
This study aims to examine the effects of mindfulness practice administered using a mobile app on psychological health among health care workers in Singapore.

DETAILED DESCRIPTION:
Research has shown that health workers are particularly at risk of experiencing heightened risks of burnout and psychological symptoms when dealing with a health pandemic, including the current COVID-19 pandemic (Lai et al., 2020; Tan et al., 2020; Wu et al., 2009). The increased risk reflects an urgent need to develop feasible psychological interventions to mitigate burnout and psychological symptoms among health workers. The present study aims to examine the effects of a brief mindfulness intervention delivered using a mobile application (HeadSpace) on psychological functioning in the context of coping with the COVID-19 pandemic in a sample of health workers in Singapore. A total of 80 health workers will be recruited and randomly assigned to using a mindfulness practice app or a cognitive games app daily over a period of 21 days. They will be assessed at baseline, post-intervention, and at one-month follow-up on depressive symptoms, anxiety, stress, burnout, compassion fatigue, compassion satisfaction, post-traumatic stress symptoms, trait mindfulness, self-compassion, sleep quality, working memory, and fear of COVID-19 infection. Results of the study will have implications on developing cost-effective interventions to mitigate psychological symptoms among health workers in the context of heightened pandemic-related stress.

ELIGIBILITY:
Inclusion Criteria:

* aged between 21 and 60
* being a health care worker based in Singapore
* proficient in English
* owns a smartphone (iOS or Android) with Wi-Fi or data access.

Exclusion Criteria:

-Regular mindfulness practice, defined by practicing a minimum of two to three times a week for 10 to 15 minutes each time within the past six months.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Depression | Change from Baseline to Within 7 Days Post intervention
  Depression subscale of the Depression, Anxiety, and Stress Scales- 21 (DASS)
Anxiety | Change from Baseline to Within 7 Days Post intervention
  Anxiety subscale of the Depression, Anxiety, and Stress Scales- 21 (DASS)
Fear of COVID-19 | Change from Baseline to Within 7 Days Post intervention
  Fear of COVID-19 Scale
Burnout, Compassion Satisfaction, and Secondary Traumatic Stress | Change from Baseline to Within 7 Days Post intervention
  Professional Quality of Life Scale Version 5 (3 subscales respectively)
Sleep Quality | Change from Baseline to Within 7 Days Post intervention
  One item from Pittsburg Sleep Quality Inventory
Working Memory | Change from Baseline to Within 7 Days Post intervention
  Digit span tasks - forward and backward
PTSD symptoms | Change from Baseline to Within 7 Days Post intervention
  Posttraumatic stress disorder Checklist- Civilian Version(higher scores indicate greater PTSD symptoms)

SECONDARY OUTCOMES:
Trait Mindfulness | Change from Baseline to Within 7 Days Post intervention
  Five Facet Mindfulness Questionnaire (higher scores indicate greater trait mindfulness)
Self-Compassion | Change from Baseline to Within 7 Days Post intervention
  Self-Compassion Scale (higher scores indicate greater self-compassion)

CONTACTS AND LOCATIONS:
Overall Officials: Shian-Ling Keng, PhD, Principal Investigator — Yale-NUS College
Locations (1):
- Yle-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keng SL, Chin JWE, Mammadova M, Teo I. Effects of Mobile App-Based Mindfulness Practice on Healthcare Workers: a Randomized Active Controlled Trial. Mindfulness (N Y). 2022;13(11):2691-2704. doi: 10.1007/s12671-022-01975-8. Epub 2022 Sep 16. PMID 36160038